CLINICAL TRIAL: NCT05485727
Title: Uses of Robotic Constraint Lokomat Training on Gait Rehabilitation in Saudi Females Patients with Stroke- a Randomized Controlled Study
Brief Title: Robotic Constraint Lokomat Training for Gait Rehabilitation in Patients with Stroke
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Umm Al-Qura University (Other)
Responsible Party: Principal Investigator, Hayam Mahmoud Sayed Mahmoud, Professor of Physical Therapy-Faculty of applied Medical Science- Physical Therapy Department, Umm Al-Qura University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Other
Other Study IDs: (HAPO-02-K-012-2022-03-1024)
Record Dates: First submitted 2022-08-01; First posted 2022-08-03 (Actual); Last update posted 2025-02-03 (Actual); Status verified 2022-08

CONDITIONS: PHYSICAL THERAPY TECHNIQUES
Keywords: Stroke, Gait, Balance, Lokomat.
MeSH Terms: conditions — Stroke

STUDY DESIGN:
Intervention Model Description: stroke patients(28) will be enrolled in this thesis (6-12 months after stroke); the Patients will be randomly assigned into two equal groups of 14. Robotic-assisted gait training group (RG) will receive Lokomat gait training and conventional physiotherapy, while the other group is a control group (CG) will receive conventional physiotherapy.
Who Masked: Outcomes Assessor
Masking Description: The outcomes assessors will not aware about the treatment procedures the participants had received before. The assessors also will be blinded about both groups( Treatment group or Control group)
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- RG(Robotic group= study group) (Experimental): 14, Robotic-assisted gait training group (RG) will receive Lokomat gait training and conventional physiotherapy
  Interventions: Other: The Lokomat® Pro Hocoma USA & Conventional physical therapy; Other: Conventional Physical Therapy
- & CG( Control group) (Active Comparator): control group (CG) will only receive conventional physiotherapy
  Interventions: Other: Conventional Physical Therapy

INTERVENTIONS:
Other: The Lokomat® Pro Hocoma USA & Conventional physical therapy — Lokomat Consists of robotic gait orthosis and an advanced body weight support system, combined with a Treadmill. (used for gait training) and Conventional Physical Therapy
  Other Names: Robotic Constraint Lokomat Training; (Enhanced Functional Locomotion Therapy with Augmented Performance Feedback)
  Arms: RG(Robotic group= study group)
Other: Conventional Physical Therapy — Balance Exercises , Gait training, Trunk control, Range of motion exercises for lower limbs
  Other Names: Designed Program of physical therapy rehabilitation for stroke patients for lower limbs

SUMMARY:
The aim of this study is to investigate the effect of a lokomat training on gait performance in Saudi females with stroke. Design: A-Single blind randomized controlled trial. Methods: 28 females patients with stroke will be enrolled in this thesis (6-12 months after stroke); the patients will be randomly assigned into two equal groups of 14. Robotic-assisted gait training group (RG) will receive Lokomat gait training and conventional physiotherapy, while the other group is a control group (CG) will receive conventional physiotherapy. Duration of treatment will be 3 months. The lower limb joint range of motion, Balance, activities of daily living, walk speed, muscle tone of the lower limbs will be recorded before and after treatment and will compared between both groups.

DETAILED DESCRIPTION:
Background: Stroke is considered one of the main causes of morbidity and mortality and the contributing cause of disability in human adults. Gait performances were dramatically affected and reduced after stroke. Purpose: The aim of this study is to investigate the effect of a lokomat training on gait performance in stroke patients of Saudi women. Design: A-Single blind randomized controlled trial. Methods: Twenty-eight females of stroke patients will be enrolled in this thesis (6-12 months after stroke); the patients will be randomly assigned into two equal groups of 14. Robotic-assisted gait training group (RG) will receive Lokomat gait training and conventional physiotherapy, while the other group is a control group (CG) will receive conventional physiotherapy. Duration of treatment will be of three months. Randomization was performed by random number generator of the Microsoft Office Excel Software. Intervention: Both groups will be evaluated before and after treatment (3-month duration). LokomatPro is designed to improve training efficiency, RG will be compared with conventional manually assisted therapy CG. The device has all the necessary elements to enable effective robotic gait training. On a treadmill, the Lokomat's powered robotic gait orthosis legs lead the subject through walking movements, supporting their body weight(with safe belts) and allowing them to use their legs more freely. Over time, the degree of body weight support and direction will be reduced to more closely resemble typical unsupported walking. The Lokomat is linked to a video game that provides feedback on the amount of force the subject will generate. The motions of the joint's angles and linear motion for lower limb (hip, knee, and ankle excursions) and Lokomat will be recorded when the patients walk on a treadmill and inside the Lokomat. Patients will walk for roughly 30 minutes three times a week for a total of twelve weeks. Instrumentations:3D Motion analysis system, with 10 cameras Bonita Model, connected with 2-force plate (AMTI), and EMG (8Channels), Nexus Version 2.5 (will used for gait analysis before and after use of lokomat). The Lokomat® Pro Hocoma USA (Enhanced Functional Locomotion Therapy with Augmented Performance Feedback) consists of the robotic gait orthosis and an advanced body weight support system, combined with a Treadmill. (used for gait training). Berg's Balance Scale (BBS) to measure balance. Modified Barthel Index (MBI) to measure activities of daily living, respectively, The Rivermead Mobility Index (RMI) will be used to assess the functional mobility of the patients (This 15-item test is a hierarchical mobility scale including rolling in bed to running, a higher score indicates better mobility performance), Modified Ashowrth Scale (MAS) For muscle tone assessment (Spasticity), Timed-Up and Go test (TUG) will be used to assess balance and functional mobility together, (a lower duration indicates better mobility performance). Outcome measure The lower limb joint range of motion, Balance, and activities of daily living, walk speed, muscle tone of the lower limbs will be recorded before and after treatment and will compared between both groups. Statistical analysis: Data calculated by using the computer package SPSS 8.0. Individual data will be expressed in mean and standard deviation (SD). Un Paired t-test will used to compare between the results of the same group before and after treatment. Paired t-test will used to compare between the results both groups after treatment with level of significance at P≤ 0.05.

ELIGIBILITY:
Inclusion Criteria:

* 28 stroke female patients, age ranged from 40- 65 years, Lower limb mild to moderate spasticity (Modified Ashwarth Scale 1+ to 3), be able to understand all instructions during intervention (Mini-Mental State Examination Score ≥24 points), & be able to walk 10 m independently or under supervision

Exclusion Criteria:

* cognitive impairment, behavioral disturbance, serious independent chronic disease likely to interfere with the ability to cooperate with the study, major contracture affecting muscles of the leg, Joint pathology of the lower limb other than that directly related to hemiplegia (eg, previous fractures, severe articular blocks); Patients under antispastic drug. Heart failure, unstable angina, uncontrolled hypertension peripheral arteriovenous occlusive disease. Neurogenic condition (other than stroke) affecting the gait pattern (e.g. ataxia, peripheral neuropathy, vertebrobasilar insufficiency and myelopathy), and patients with advanced osteoarthritis, and obesity (BMI > 30)

Ages: 40 Years to 65 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes — 28 females of stroke patients will be enrolled in this thesis (6-12 months after stroke); the patients will be randomly assigned into two equal groups of 14.
Enrollment: 28 (Actual)
Dates: Start 2022-03-30 (Actual); Primary Completion 2023-09-30 (Actual); Study Completion 2023-12-10 (Actual)

PRIMARY OUTCOMES:
lower limb joint range of motion | 3 months
  3D Motion analysis system, with 10 cameras Bonita Model, connected with 2-force plate (AMTI), and EMG (8Channels), Nexus Version 2.5 (will used for gait analysis before and after lokomat usage)
Balance | 3 months
  Berg's Balance Scale (BBS) to measure balance
Activities of daily living | 3 months
  Modified Barthel Index (MBI) to measure activities of daily living
Spasticity of the lower limbs | 3 months
  Modified Ashowrth Scale (MAS) For muscle tone assessment (Spasticity
Gait speed | 3 months
  Timed-Up and Go test (TUG) will be used to assess gait speed with dynamic balance

CONTACTS AND LOCATIONS:
Overall Officials: Hayam Mahmoud, professor, Principal Investigator — Umm Al-Qura University
Locations (2):
- Saudi Arabia (2):
  - Faculty of Applied Medical Science - UQU, Jeddah
  - UQU- KSA, Jeddah

IPD SHARING:
Plan to Share IPD: Yes
Results , Methodology , Publication
Supporting Information: Study Protocol, SAP, ICF, Analytic Code
Time Frame: One year
Access Criteria: Published article, or paper

REFERENCES:
- [Derived] Mahmoud H, El-Kafy EA, Alayat MS, Shalabi KM, Ebid AA, El Fiky AAR. The Effectiveness of Robotic Constraint Lokomat Training on Gait Rehabilitation in Saudi Females Patients with Stroke: A Randomized Controlled Trial. NeuroRehabilitation. 2025 Aug;57(1):70-79. doi: 10.1177/10538135251333349. Epub 2025 May 11. PMID 40350663